CLINICAL TRIAL: NCT04196998
Title: Study on Therapeutic Effects and Safety of Three Types of Nucleotide/Nucleoside Analogues in Patients With Hepatitis b Virus Related Compensated Cirrhosis
Brief Title: Three Types of Nucleotide/Nucleoside Analogues Therapy in Patients With Hepatitis b Virus Related Compensated Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professer, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XWX2
Record Dates: First submitted 2019-12-09; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis B; Compensated Cirrhosis
Keywords: hepatitis b virus; compensated cirrhosis; nucleoside; nucleotide
MeSH Terms: conditions — Hepatitis B | interventions — entecavir; Tenofovir; tenofovir alafenamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ETV group (Active Comparator): 50 patients would receive treatment of oral entecavir (ETV) 0.5 mg once per day from baseline to life-long.
  Interventions: Drug: Entecavir
- TDF group (Active Comparator): 50 patients would receive treatment of oral tenofovir disoproxil fumarate (TDF) 300 mg once per day from baseline to life-long.
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- TAF group (Experimental): 50 patients would receive treatment of oral tenofovir alafenamide (TAF) 25 mg once per day from baseline to life-long.
  Interventions: Drug: Tenofovir alafenamide

INTERVENTIONS:
Drug: Entecavir — Patients would receive treatment of oral entecavir (ETV) 0.5 mg once per day.
  Other Names: Baraclude
  Arms: ETV group
Drug: Tenofovir Disoproxil Fumarate — Patients would receive treatment of oral tenofovir disoproxil fumarate (TDF) 300 mg once per day.
  Other Names: Viread
  Arms: TDF group
Drug: Tenofovir alafenamide — Patients would receive treatment of oral tenofovir alafenamide (TAF) 25 mg once per day.
  Other Names: Vemlidy
  Arms: TAF group

SUMMARY:
This study is to investigate the clinical efficacy and safety of three types of nucleotide/nucleoside analogues in treatment of hepatitis b virus related compensated cirrhosis.

DETAILED DESCRIPTION:
Hepatitis b virus infection remains a serious public health problem in China. Nucleotide/nucleoside analogues are used for anti-virus treatment in these patients. Entecavir, Tenofovir Disoproxil Fumarate and Tenofovir Alafenamide are first line drug in China. But there still lacks of data of Tenofovir Alafenamide in treatment of hepatitis b virus related compensated cirrhosis. This study is to investigate the clinical efficacy and safety of three types of nucleotide/nucleoside analogues in treatment of hepatitis b virus related compensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Positive hepatitis b surface antigen or hepatitis b virus DNA > 0.5 year;
2. Age from 18 to 65 years old;
3. Hepatitis b virus DNA positive;
4. Cirrhosis or portal hypertension is found through ultrasonography, computed tomography or magnetic resonance imaging;
5. Do not receive nucleotide/nucleoside analogues treatment in the past half year.

Exclusion Criteria:

1. Complications of decompensated cirrhosis: ascites, gastrointestinal bleeding, hepatic encephalopathy, hepatorenal syndrome, etc;
2. Other active liver diseases;
3. Hepatocellular carcinoma or other malignancy;
4. Pregnancy or lactation;
5. Human immunodeficiency virus infection or congenital immune deficiency diseases;
6. Severe diabetes, autoimmune diseases;
7. Other important organ dysfunctions;
8. Using glucocorticoid;
9. Patients can not follow-up;
10. Investigator considering inappropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of decompensated cirrhosis | 144 week
  Incidence of decompensated cirrhosis is evaluated in the follow-up

SECONDARY OUTCOMES:
Ratio of patients with undetectable hepatitis b virus DNA after treatment | 4 week, 8 week, 12 week, 24 week, 48 week, 72 week,144 week
  Hepatitis b virus DNA would be tested to know the ratio of patients with undetectable hepatitis b virus DNA at 7 time points after treatment.
Ratio of patients with hepatitis b virus e antigen seroconversion after treatment | 4 week, 8 week, 12 week, 24 week, 48 week, 72 week,144 week
  Hepatitis b virus e antigen and e antibody would be tested to know the ratio of patients with hepatitis b virus e antigen seroconversion at 7 time points after treatment.
Ratio of patients with undetectable hepatitis b virus surface antigen after treatment | 4 week, 8 week, 12 week, 24 week, 48 week, 72 week,144 week
  Hepatitis b virus surface antigen would be tested to know the ratio of patients with undetectable hepatitis b virus surface antigen at 7 time points after treatment.
Serum calcium | 4 week, 8 week, 12 week, 24 week, 48 week, 72 week,144 week
  Hypocalcemia would be evaluated after treatment
Serum phosphorus | 4 week, 8 week, 12 week, 24 week, 48 week, 72 week,144 week
  Hypophosphatemia would be evaluated after treatment
Blood urea nitrogen | 4 week, 8 week, 12 week, 24 week, 48 week, 72 week,144 week
  Blood urea nitrogen would be tested after treatment
Serum creatinine | 4 week, 8 week, 12 week, 24 week, 48 week, 72 week,144 week
  Serum creatinine would be tested after treatment
Estimated glomerular filtration rate | 4 week, 8 week, 12 week, 24 week, 48 week, 72 week,144 week
  Estimated glomerular filtration rate would be evaluated after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China